CLINICAL TRIAL: NCT04443452
Title: Molecular Pathways Involved in Knee Pain: an Observational Study
Brief Title: Molecular Pathways Involved in Knee Pain
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Versus Arthritis (Other)
Responsible Party: Sponsor
Other Study IDs: 19098; 22473 (Other Grant/Funding Number: Versus Arthritis); 275727 (Other: IRAS)
Record Dates: First submitted 2020-06-05; First posted 2020-06-23 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-04

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Postsynaptic Potential Summation; X-Rays; Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Saliva, Synovial fluid from the most painful knee, Faeces (OPTIONAL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prevalent Central Sensitisation: Participants with sensitisation that significantly deviates from the normal mean as assessed by Quantitative Sensory Testing
  Interventions: Diagnostic Test: Quantitative Sensory Testing; Radiation: Radiographic Evaluation; Procedure: Ultrasound-guided Aspiration; Diagnostic Test: Muscle Strength Assessment; Diagnostic Test: Function Assessment (A); Diagnostic Test: Function Assessment (B); Diagnostic Test: Balance Assessment
- Non-prevalent Central Sensitisation: All other participants with sensitisation that is not significantly deviating from the normal mean as assessed by Quantitative Sensory Testing
  Interventions: Diagnostic Test: Quantitative Sensory Testing; Radiation: Radiographic Evaluation; Procedure: Ultrasound-guided Aspiration; Diagnostic Test: Muscle Strength Assessment; Diagnostic Test: Function Assessment (A); Diagnostic Test: Function Assessment (B); Diagnostic Test: Balance Assessment

INTERVENTIONS:
Diagnostic Test: Quantitative Sensory Testing — PPT: An electronic data collection unit will be used featuring an electronic algometer connected with a laptop where the amount of pressure will be displayed on the screen. When the pressure pain detection threshold is reached (the point where the pressure sensation starts to be experienced as pain), the individual will press a button at a handheld device, that will automatically store the pressure value in the system and serve as an indication, for the examiner, to stop the testing.
  TS: A pinprick stimulator (Weight: 256mNewton) will be used. The examiner will apply the pen that features a retractable blunt needle in a repetitive manner (once per second for ten seconds). The individual will be asked for the intensity of pain (NRS) at the first and at the last time and the given score will be noted.
  CPM: A manual blood pressure sphygmomanometer will be used in conjunction with the electronic algometer described above (PPT).
  Other Names: Pressure Pain Detection Threshold (PPT); Temporal Summation (TS); Conditioned Pain Modulation (CPM)
Radiation: Radiographic Evaluation — Tibiofemoral and patellofemoral radiographs of the most painful knee will be taken using a standardised protocol (standing posterior-anterior (PA) and skyline views) and will be scored by a single experienced observer in order to generate data for correlation analyses with the primary and secondary outcomes. A Perspex Rosenberg template with lead beads is used for the standing PA view to standardising the degree of knee flexion, foot rotation and magnification. PA radiographs are taken with the participant facing the x-ray tube while standing on the Rosenberg jig and leaning forwards with their thighs touching the anterior aspect of the jig, the x-ray beams passing from the posterior aspect through to the anterior aspect of the knee. Variable jigs are used for the skyline view to obtaining 300 of knee flexion with the participant lying in a reclined supine position on a couch. Grading of radiographs for changes of OA will be based on the Kellgren and Lawrence (K/L) score.
  Other Names: X-rays
Procedure: Ultrasound-guided Aspiration — Ultrasound scanning will be conducted on the most painful knee to identify synovial effusion. During the ultrasound scan, the supra-patellar pouch, medial and lateral recess of the knees will be assessed for synovial thickening, synovial fluid/effusion and for positive power Doppler. An ultrasonic probe will be used to direct ultrasonic waves onto the knee joint during sonography, and a computer converts the signals received so that they can be presented on the screen. During skin application, a sterile probe cover and sterile acoustic gel will be used. Once the best aspiration location is identified and the location of the needle insertion marked, the skin will be prepared with a cleansing agent such as iodine or chlorhexidine. The needle may be introduced into the skin either parallel to the probe or perpendicular to the probe. Once the aspiration is completed, the needle will be removed, the skin cleansed, and a bandage will be applied.
  Other Names: Synovial Fluid Extraction
Diagnostic Test: Muscle Strength Assessment — Isometric testing will be done at 30 and 60 degrees of flexion as done in the previous study and the participant will be in sitting position with hips and knees strapped to keep the position standardised.
  Other Names: Isometric Dynamometer
Diagnostic Test: Function Assessment (A) — The participant will start in a seated position. The participant will stand up upon therapist's command, walk 3 meters, turn around, walk back to the chair and sit down. The time will stop when the participant is seated. The subject can use an assistive device. If the assistive device is used, it will be documented.
  Important Note: A practice trial will be completed before the timed trial.
  Other Names: Time Up-and-Go Test
Diagnostic Test: Function Assessment (B) — The 30-Second Chair Test is administered using a chair. The participant is seated in the middle of the chair with arms crossed at the wrists and held against the chest. The participant will practice a repetition or 2 before completing the test. If a participant must use their arms to complete the test, they are scored 0. The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand. While monitoring the participant's performance to ensure proper form, the tester silently counts the completion of each correct stand. The score is the total number of stands within 30 seconds (more than halfway up at the end of 30 seconds counts as a full stand). Incorrectly executed stands are not counted. The 30-second chair stand involves recording the number of stands a person can complete in 30 seconds rather than the amount of time it takes to complete a pre-determined number of repetitions.
  Other Names: 30 seconds Sit-to-Stand Test
Diagnostic Test: Balance Assessment — Static balance and postural sway either in the medial-lateral or antero-posterior direction will be assessed using the RS Scan force plate. The participant will be asked to stand on the plate looking straight forward for 30 seconds in two conditions: first with their eyes open and then with eyes closed. Medial-lateral, antero-posterior and total sway will be recorded.
  Other Names: Static Balance Test; Postural Sway Test

SUMMARY:
Knee osteoarthritis (OA) is the most common form of arthritis and the most common cause of knee pain in the world. The rate of knee arthritis is as high as that of cardiac disease and is the most common problem in individuals over the age of 65.

Central Sensitization (CS) is a marker of widespread pain sensitivity that can occur throughout the central nervous system distribution, leading to changes in the spinal cord as well as in the brain. The presence of CS increases the complexity of the clinical picture and can negatively affect treatment outcomes. CS is present in >20% of patients suffering from knee OA indicating that in the majority of individuals suffering with painful knee OA, knee pain should be related to molecular changes in the joint. CS might be also associated with discrete synovial fluid proteomic signatures due to the generation by the joint of chemical mediators (e.g. nerve growth factor) that drive CS, or CS might moderate the relationship between synovial fluid proteomic signatures and symptoms due to alterations in pain processing.

The aim of this study is to explore the potential molecular links between pain and structure on knee pain using synovial fluid proteomics. A secondary purpose is to explore the association of knee pain with biomarkers of stress, metabolism and dietary habits.

In a single session, ultrasound-guided synovial fluid, blood urine and saliva extraction, clinical assessment, completion of a questionnaire booklet and knee x-rays will be conducted. The clinical assessment will measure three features of central sensitisation (sensitivity to blunt pressure on the most painful knee, changes in pain felt during repeated light pricking of the knee skin, and reduction in pain that accompanies inflation of a blood pressure cuff on the non-dominant arm), features of leg strength (dynamometer, time up-and-go test) and features of balance (sway). Participant involvement at each session is expected to last less than 3 hours.

Individuals over 45 having complaints of knee pain for 3-6 months are eligible to participate. The clinical assessments, questionnaire completion and subsequent statistical analysis are expected to be completed within 18 months of study commencement.

The findings can provide more insight into the traits of knee pain, allow the examination of possible correlations to each other, and highlight potential detrimental effects of them on knee joint health.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common cause of disability in the elderly population and most individuals suffering from osteoarthritis are managed in the primary care setting. Knee OA is the most common form of arthritis and the most common cause of knee pain in the world. The rate of knee arthritis is as high as that of cardiac disease and is the most common problem in individuals over the age of 65. In the United Kingdom, 10% of 65 to 74-year-old individuals consult their general practitioners about OA per year. Out of the entire population, 4% attend their general practitioners as a result of knee OA, and half of them (2%) consult their general practitioner for the first time or with the acute flare of knee arthritis.

There is a considerable body of evidence showing augmented central nervous system (CNS) processing in OA. Central Sensitization (CS) is a marker of widespread and centrally augmented pain that refers to those neurophysiological processes that can occur throughout the CNS distribution, leading to changes in the spinal cord as well as in the brain. The presence of CS increases the complexity of the clinical picture and negatively affects a range of outcomes (e.g. pain, disability, negative affect, quality of life) following treatment. CS is not present within all patients with chronic pain rendering identification of those patients and decision-making for the right management approach even harder. Clinically, CS manifests as hypersensitivity to pain, that sometimes spreads beyond peripheral generators and is a marker for pain chronicity. CS of nociceptive pathways is a mechanism of clinical pain amplification in OA and is present in >20% of patients suffering from knee OA. This means that in the majority of individuals suffering with painful knee OA, knee pain should be related to molecular changes in the joint. CS might be also associated with discrete synovial fluid proteomic signatures due to the generation by the joint of chemical mediators (e.g. nerve growth factor) that drive CS, or CS might moderate the relationship between synovial fluid proteomic signatures and symptoms due to alterations in pain processing. Radiographic knee joint changes and pain levels are associated with knee cartilage loss but whether CS indices are linked to radiographic changes has not been established. High levels of CS might increase the risk of cartilage loss by increasing the levels of pain or might be associated with already existing changes.

The investigators will recruit 140 individuals with OA-related knee pain. They will also use standardised quantitative sensory testing (QST) such as pressure pain detection threshold (PPT), temporal summation (TS) and conditioned pain modulation (CPM). PPT specifically, has been used in past knee pain studies and is considered a valid and reliable method to establish tenderness around the knee joint. Similarly, TS has been used previously to establish whether individuals demonstrate amplified, centrally driven localised knee pain. Conditioned pain paradigms are commonly used to assess the function of endogenous pain inhibitory pathways in humans. In this technique, a painful test stimulus is evaluated in the absence and then in the presence of a second, also painful (conditioning), stimulus applied to a remote region of the body. In a typically functioning nociceptive system, the amount of pain experienced with the primary test stimulus will be reduced during the presentation of the secondary conditioning stimulus. Decreased inhibition of experimental pain is found in many patients with idiopathic pain syndromes. It predicts the tendency to develop future chronic pain. The purpose of using QST is to establish objective and quantifiable data that will allow the stratification of patients into 'sensitised' and 'non-sensitised' and permit further analysis.

Quantitative Sensory Testing is a reliable and valid method to assess for the presence of CS and demonstrates predictive capacity in relation to musculoskeletal (MSK) treatment outcomes. The testing consists of pressure pain threshold (PPT), punctate thresholds, temperature sensitivity, temporal summation (TS) and conditioned pain modulation (CPM) used to quantify noxious or innocuous stimuli within healthy individuals and patients alike. QST has been used, among others, as a screening and assessment tool for sensory abnormalities in patients with pain disorders, as well as to assist in the stratification of patients and evaluate the clinical aspects of peripheral and CS.

Regional pain and symptoms of depression and/or anxiety have been shown to facilitate the development of constant pain therefore, signs of depression or anxiety are important to explore correlation of symptoms at a single time-point. Signs of depression and anxiety can be identified with the use of the Hospital Anxiety and Depression Scale (HADS) that has been shown to be valid in multiple populations. The stress response involves activation of the sympathetic nervous system and the hypothalamic-pituitary-adrenal (HPA) axis. Any physical or psychological threat to homeostasis triggers release of corticotrophin-releasing hormone in the hypothalamus, and ultimately raises levels of steroid hormones such as cortisol in the blood stream and saliva. In the short term, cortisol helps to meet the demands of stress by mobilizing energy stores, and assists recovery from stress by inhibiting further release of corticotrophin-releasing hormone. However, continuing stress promotes maladaptive functioning of the HPA axis, which, in turn, may compromise metabolism, impair immune function, and alter cardiovascular control. Cortisol levels in saliva have been implicated in chronic pain presentations (pain severity) and can be considered a useful biological biomarker that can be used to explore psychopathological associations, prognosis and treatment outcomes.

Nutritional information collected via a standardised food frequency questionnaire (FFQ) and metabolic evidence from body secretions can provide significant insight about the course of OA, as the presence of glucosamine and chondroitin sulfate in faecal samples has shown to improve the symptoms of the condition and delay its progression. Nutritional information and metabolic evidence from faecal samples can be used to explore associations of gut microbiota with pain sensitivity and stress levels.

The widely utilised Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) will be also used for the evaluation of knee OA. It is a self-administered questionnaire made of 24 items and consists of three subscales covering pain, stiffness and physical function. It has been used extensively and is considered a valid and reliable tool. For evaluating quality of life, stiffness, generalised well-being, sleeping difficulties and understanding of the diagnosis and treatment, the investigators will use patient-reported outcome measure 'The Versus Arthritis Musculoskeletal Health Questionnaire' (MSK-HQ). MSK-HQ covers a broad aspect of musculoskeletal conditions, and recent studies have shown it to be reliable and valid. Frailty has been also found to be a predictor of disability and a determinant of treatment outcomes and the Simple Frailty Questionnaire (FRAIL) is considered a valid and reliable tool for that purpose.

Both the 30-second sit to stand test (30CST) and the 'time up and go' (TUG) test will be used to see if patients have improved their lower limb fitness levels. 30CST has shown excellent reliability and validity. TUG has been widely used in clinical setups and is a valid tool to assess necessary functional mobility.

In this study, the sleeping pattern of individuals suffering from degenerative changes of the knee will be assessed with the aim to establish whether sleep disturbance is implicated in the development of CS. Disturbed sleep is a frequent complaint of people experiencing chronic pain such as those with knee osteoarthritis (OA). Changes in sleep architecture can affect health even in the presence of apparently adequate sleep duration. Insufficient amounts of slow wave sleep are associated with hypertension, type 2 diabetes mellitus, poor cognition, and obesity. Sleep disturbances are present in 67-88% of people with chronic pain and ≥50% individuals with insomnia have chronic pain. The investigators will also use the Pittsburgh sleep quality index (PSQI) which has been used in multiple studies and validated to measure sleep disturbances. Poor cognition, as well as sleep, has been found to be a marker of persistent pain and a trait of centrally driven pain in knee pain populations. The Cognitive Failures Questionnaire (CFQ) is a valid and reliable tool to measure self-reported failures in perception, memory, and motor function.

Musculoskeletal Ultrasound scan (MSK-USS) will be also conducted on the knees of participants to establish if they have inflammation of the synovial membrane. There is enough evidence that inflammation is present in all stages of OA. Synovitis or inflammation of synovial fluid is associated with pain, disease severity and, OA progression. Synovitis manifests as synovial membrane thickening, increased vascularity, and/or joint effusion. Synovial hypertrophy, synovitis and knee effusion are linked with arthritis in the knee and associated with knee pain in osteoarthritis. The synovial fluid will be aspirated (subject to participant consent), in order to establish a phenotype which is strongly associated with OA. Studying synovial fluid biomarkers alongside clinical, radiographic and ultra-sonographic characteristics is one strategy to improve resolution and stratification into targetable OA phenotypes. Synovial fluid aspiration will be ultrasound guided as it increases the accuracy of needle placement compared to blind needling (95.8% versus 77.8%, p < 0.001) reduces procedural pain by 43%, improves effusion detection by 200%, and volume of synovial fluid aspirated by 337% compared with blind synovial fluid aspiration. Ultrasound guidance also reduces procedural pain (43% reduction) in knees with no palpable effusion and increases the responder rate and therapeutic duration by 107% and 36% respectively.

Isometric quadriceps strength will be also assessed to establish current strength levels of vastus medialis muscle and see whether muscle strength associates with centrally driven pain or proteomic synovial concentrations. Quadriceps muscles strength deficits are associated with knee osteoarthritis. Isometric testing will be done at 30 and 60 degrees of flexion as per the protocol of a previous study.

Blood samples will be also extracted to assess the biomarkers (including serum levels and gene expression levels of various molecules) and to establish insulin resistance. Urine samples will be collected to identify the existence of collagen degradation markers (e.g. UTXII) and inflammatory regulator markers (e.g. Maresins).

Collection and study of these parameters can provide more insight into the traits of knee pain, allow the examination of possible correlations to each other, and highlight potential detrimental effects of them on knee joint health.

ELIGIBILITY:
Inclusion Criteria:

* have the ability to give informed consent
* be 45 years or over
* have complaints of knee pain for 3-6 months with or without radiographically established OA (K/L scale score ≥ 1)
* have complaints of knee pain for 3-6 months with or without satisfying the non-radiographic American College of Rheumatology criteria for knee OA
* are willing to undertake knee synovial fluid aspiration
* be able to speak, read, and write in English as all instructions and questionnaires are designed in the English language

Exclusion Criteria:

* Inability to give informed consent due to cognitive impairment or otherwise - (capacity levels are already established under General Practitioner care)
* Inability to understand key aspects of the study due to cognitive impairment or otherwise
* Giving history of additional co-morbidities such as cancer, neurological conditions, inflammatory joint diseases including rheumatoid arthritis, diabetic neuropathies, fractures or other conditions causing greater disability than their knee pain
* Acute soft tissue injury to the knee within last 3 months before potential recruitment

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults equal or above the age of 45 with a history of knee pain of at least 3 months duration that may or may not have been radiographically and no-radiographically classified as having knee pain due to osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Valdes, PhD, Principal Investigator — University of Nottingham
Locations (1):
- The University of Nottingham, City Hospital Campus, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Considerations about data sharing will be taken once the main results of this study have been published

REFERENCES:
- [Background] Peat G, McCarney R, Croft P. Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Ann Rheum Dis. 2001 Feb;60(2):91-7. doi: 10.1136/ard.60.2.91. PMID 11156538
- [Background] Felson DT. Weight and osteoarthritis. Am J Clin Nutr. 1996 Mar;63(3 Suppl):430S-432S. doi: 10.1093/ajcn/63.3.430. PMID 8615335
- [Background] Guccione AA, Felson DT, Anderson JJ, Anthony JM, Zhang Y, Wilson PW, Kelly-Hayes M, Wolf PA, Kreger BE, Kannel WB. The effects of specific medical conditions on the functional limitations of elders in the Framingham Study. Am J Public Health. 1994 Mar;84(3):351-8. doi: 10.2105/ajph.84.3.351. PMID 8129049
- [Background] McCormick, A. Morbidity statistics from general practice. Fourth national study 1991-1992. Office of population censuses and surveys.1995.
- [Background] Finan PH, Buenaver LF, Bounds SC, Hussain S, Park RJ, Haque UJ, Campbell CM, Haythornthwaite JA, Edwards RR, Smith MT. Discordance between pain and radiographic severity in knee osteoarthritis: findings from quantitative sensory testing of central sensitization. Arthritis Rheum. 2013 Feb;65(2):363-72. doi: 10.1002/art.34646. PMID 22961435
- [Background] Malfait AM, Schnitzer TJ. Towards a mechanism-based approach to pain management in osteoarthritis. Nat Rev Rheumatol. 2013 Nov;9(11):654-64. doi: 10.1038/nrrheum.2013.138. Epub 2013 Sep 17. PMID 24045707
- [Background] Latremoliere A, Woolf CJ. Central sensitization: a generator of pain hypersensitivity by central neural plasticity. J Pain. 2009 Sep;10(9):895-926. doi: 10.1016/j.jpain.2009.06.012. PMID 19712899
- [Background] Nijs J, Van Oosterwijck J, De Hertogh W. Rehabilitation of chronic whiplash: treatment of cervical dysfunctions or chronic pain syndrome? Clin Rheumatol. 2009 Mar;28(3):243-51. doi: 10.1007/s10067-008-1083-x. Epub 2009 Jan 22. PMID 19160000
- [Background] Jull G, Sterling M, Kenardy J, Beller E. Does the presence of sensory hypersensitivity influence outcomes of physical rehabilitation for chronic whiplash?--A preliminary RCT. Pain. 2007 May;129(1-2):28-34. doi: 10.1016/j.pain.2006.09.030. Epub 2007 Jan 10. PMID 17218057
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Murphy SL, Lyden AK, Phillips K, Clauw DJ, Williams DA. Subgroups of older adults with osteoarthritis based upon differing comorbid symptom presentations and potential underlying pain mechanisms. Arthritis Res Ther. 2011 Aug 24;13(4):R135. doi: 10.1186/ar3449. PMID 21864381
- [Background] French HP, Smart KM, Doyle F. Prevalence of neuropathic pain in knee or hip osteoarthritis: A systematic review and meta-analysis. Semin Arthritis Rheum. 2017 Aug;47(1):1-8. doi: 10.1016/j.semarthrit.2017.02.008. Epub 2017 Feb 20. PMID 28320529
- [Background] Saunders J, Ding C, Cicuttini F, Jones G. Radiographic osteoarthritis and pain are independent predictors of knee cartilage loss: a prospective study. Intern Med J. 2012 Mar;42(3):274-80. doi: 10.1111/j.1445-5994.2011.02438.x. PMID 21299779
- [Background] Geber C, Klein T, Azad S, Birklein F, Gierthmuhlen J, Huge V, Lauchart M, Nitzsche D, Stengel M, Valet M, Baron R, Maier C, Tolle T, Treede RD. Test-retest and interobserver reliability of quantitative sensory testing according to the protocol of the German Research Network on Neuropathic Pain (DFNS): a multi-centre study. Pain. 2011 Mar;152(3):548-556. doi: 10.1016/j.pain.2010.11.013. Epub 2011 Jan 14. PMID 21237569
- [Background] Pfau DB, Krumova EK, Treede RD, Baron R, Toelle T, Birklein F, Eich W, Geber C, Gerhardt A, Weiss T, Magerl W, Maier C. Quantitative sensory testing in the German Research Network on Neuropathic Pain (DFNS): reference data for the trunk and application in patients with chronic postherpetic neuralgia. Pain. 2014 May;155(5):1002-1015. doi: 10.1016/j.pain.2014.02.004. Epub 2014 Feb 10. PMID 24525274
- [Background] Sterling M, Jull G, Vicenzino B, Kenardy J, Darnell R. Physical and psychological factors predict outcome following whiplash injury. Pain. 2005 Mar;114(1-2):141-8. doi: 10.1016/j.pain.2004.12.005. Epub 2005 Jan 21. PMID 15733639
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Lee YC, Lu B, Bathon JM, Haythornthwaite JA, Smith MT, Page GG, Edwards RR. Pain sensitivity and pain reactivity in osteoarthritis. Arthritis Care Res (Hoboken). 2011 Mar;63(3):320-7. doi: 10.1002/acr.20373. Epub 2010 Oct 18. PMID 20957660
- [Background] Neogi T, Frey-Law L, Scholz J, Niu J, Arendt-Nielsen L, Woolf C, Nevitt M, Bradley L, Felson DT; Multicenter Osteoarthritis (MOST) Study. Sensitivity and sensitisation in relation to pain severity in knee osteoarthritis: trait or state? Ann Rheum Dis. 2015 Apr;74(4):682-8. doi: 10.1136/annrheumdis-2013-204191. Epub 2013 Dec 18. PMID 24351516
- [Background] Neogi T, Guermazi A, Roemer F, Nevitt MC, Scholz J, Arendt-Nielsen L, Woolf C, Niu J, Bradley LA, Quinn E, Law LF. Association of Joint Inflammation With Pain Sensitization in Knee Osteoarthritis: The Multicenter Osteoarthritis Study. Arthritis Rheumatol. 2016 Mar;68(3):654-61. doi: 10.1002/art.39488. PMID 26554395
- [Background] Wessel J. The reliability and validity of pain threshold measurements in osteoarthritis of the knee. Scand J Rheumatol. 1995;24(4):238-42. doi: 10.3109/03009749509100881. PMID 7481589
- [Background] Pud D, Granovsky Y, Yarnitsky D. The methodology of experimentally induced diffuse noxious inhibitory control (DNIC)-like effect in humans. Pain. 2009 Jul;144(1-2):16-9. doi: 10.1016/j.pain.2009.02.015. Epub 2009 Apr 8. No abstract available. PMID 19359095
- [Background] Yarnitsky D, Arendt-Nielsen L, Bouhassira D, Edwards RR, Fillingim RB, Granot M, Hansson P, Lautenbacher S, Marchand S, Wilder-Smith O. Recommendations on terminology and practice of psychophysical DNIC testing. Eur J Pain. 2010 Apr;14(4):339. doi: 10.1016/j.ejpain.2010.02.004. Epub 2010 Mar 12. No abstract available. PMID 20227310
- [Background] Lewis GN, Rice DA, McNair PJ. Conditioned pain modulation in populations with chronic pain: a systematic review and meta-analysis. J Pain. 2012 Oct;13(10):936-44. doi: 10.1016/j.jpain.2012.07.005. Epub 2012 Sep 13. PMID 22981090
- [Background] Chang L. Brain responses to visceral and somatic stimuli in irritable bowel syndrome: a central nervous system disorder? Gastroenterol Clin North Am. 2005 Jun;34(2):271-9. doi: 10.1016/j.gtc.2005.02.003. PMID 15862935
- [Background] Julien N, Goffaux P, Arsenault P, Marchand S. Widespread pain in fibromyalgia is related to a deficit of endogenous pain inhibition. Pain. 2005 Mar;114(1-2):295-302. doi: 10.1016/j.pain.2004.12.032. PMID 15733656
- [Background] Kosek E, Hansson P. Modulatory influence on somatosensory perception from vibration and heterotopic noxious conditioning stimulation (HNCS) in fibromyalgia patients and healthy subjects. Pain. 1997 Mar;70(1):41-51. doi: 10.1016/s0304-3959(96)03295-2. PMID 9106808
- [Background] Lautenbacher S, Rollman GB. Possible deficiencies of pain modulation in fibromyalgia. Clin J Pain. 1997 Sep;13(3):189-96. doi: 10.1097/00002508-199709000-00003. PMID 9303250
- [Background] Maixner W, Fillingim R, Booker D, Sigurdsson A. Sensitivity of patients with painful temporomandibular disorders to experimentally evoked pain. Pain. 1995 Dec;63(3):341-351. doi: 10.1016/0304-3959(95)00068-2. PMID 8719535
- [Background] Pielsticker A, Haag G, Zaudig M, Lautenbacher S. Impairment of pain inhibition in chronic tension-type headache. Pain. 2005 Nov;118(1-2):215-23. doi: 10.1016/j.pain.2005.08.019. Epub 2005 Oct 3. PMID 16202520
- [Background] Rossi P, Serrao M, Perrotta A, Pierelli F, Sandrini G, Nappi G. Neurophysiological approach to central pain modulation in primary headaches. J Headache Pain. 2005 Sep;6(4):191-4. doi: 10.1007/s10194-005-0182-1. PMID 16362661
- [Background] Sandrini G, Rossi P, Milanov I, Serrao M, Cecchini AP, Nappi G. Abnormal modulatory influence of diffuse noxious inhibitory controls in migraine and chronic tension-type headache patients. Cephalalgia. 2006 Jul;26(7):782-9. doi: 10.1111/j.1468-2982.2006.01130.x. PMID 16776692
- [Background] Song GH, Venkatraman V, Ho KY, Chee MW, Yeoh KG, Wilder-Smith CH. Cortical effects of anticipation and endogenous modulation of visceral pain assessed by functional brain MRI in irritable bowel syndrome patients and healthy controls. Pain. 2006 Dec 15;126(1-3):79-90. doi: 10.1016/j.pain.2006.06.017. Epub 2006 Jul 18. PMID 16846694
- [Background] Edwards RR, Ness TJ, Weigent DA, Fillingim RB. Individual differences in diffuse noxious inhibitory controls (DNIC): association with clinical variables. Pain. 2003 Dec;106(3):427-437. doi: 10.1016/j.pain.2003.09.005. PMID 14659526
- [Background] Yarnitsky D, Crispel Y, Eisenberg E, Granovsky Y, Ben-Nun A, Sprecher E, Best LA, Granot M. Prediction of chronic post-operative pain: pre-operative DNIC testing identifies patients at risk. Pain. 2008 Aug 15;138(1):22-28. doi: 10.1016/j.pain.2007.10.033. Epub 2008 Jan 8. PMID 18079062
- [Background] Soni A, Kiran A, Hart DJ, Leyland KM, Goulston L, Cooper C, Javaid MK, Spector TD, Arden NK. Prevalence of reported knee pain over twelve years in a community-based cohort. Arthritis Rheum. 2012 Apr;64(4):1145-52. doi: 10.1002/art.33434. Epub 2011 Dec 16. PMID 22180258
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Julian LJ. Measures of anxiety: State-Trait Anxiety Inventory (STAI), Beck Anxiety Inventory (BAI), and Hospital Anxiety and Depression Scale-Anxiety (HADS-A). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S467-72. doi: 10.1002/acr.20561. No abstract available. PMID 22588767
- [Background] Spinhoven P, Ormel J, Sloekers PP, Kempen GI, Speckens AE, Van Hemert AM. A validation study of the Hospital Anxiety and Depression Scale (HADS) in different groups of Dutch subjects. Psychol Med. 1997 Mar;27(2):363-70. doi: 10.1017/s0033291796004382. PMID 9089829
- [Background] Biondi M, Picardi A. Psychological stress and neuroendocrine function in humans: the last two decades of research. Psychother Psychosom. 1999;68(3):114-50. doi: 10.1159/000012323. PMID 10224513
- [Background] Spiegel D, Kato PM. Psychosocial influences on cancer incidence and progression. Harv Rev Psychiatry. 1996 May-Jun;4(1):10-26. doi: 10.3109/10673229609030518. PMID 9384968
- [Background] De Kloet ER, Derijk R. Signaling pathways in brain involved in predisposition and pathogenesis of stress-related disease: genetic and kinetic factors affecting the MR/GR balance. Ann N Y Acad Sci. 2004 Dec;1032:14-34. doi: 10.1196/annals.1314.003. PMID 15677393
- [Background] Vachon-Presseau E, Roy M, Martel MO, Caron E, Marin MF, Chen J, Albouy G, Plante I, Sullivan MJ, Lupien SJ, Rainville P. The stress model of chronic pain: evidence from basal cortisol and hippocampal structure and function in humans. Brain. 2013 Mar;136(Pt 3):815-27. doi: 10.1093/brain/aws371. PMID 23436504
- [Background] Evans KD, Douglas B, Bruce N, Drummond PD. An exploratory study of changes in salivary cortisol, depression, and pain intensity after treatment for chronic pain. Pain Medicine. 2008;9(6):752-8.
- [Background] National Institutes of Health. National Cancer Institute (2017) Dietary assessment primer, food frequency questionnaire at a glance. 2017.
- [Background] Messina OD, Vidal Wilman M, Vidal Neira LF. Nutrition, osteoarthritis and cartilage metabolism. Aging Clin Exp Res. 2019 Jun;31(6):807-813. doi: 10.1007/s40520-019-01191-w. Epub 2019 Apr 13. PMID 30982220
- [Background] De Palma G, Collins SM, Bercik P, Verdu EF. The microbiota-gut-brain axis in gastrointestinal disorders: stressed bugs, stressed brain or both? J Physiol. 2014 Jul 15;592(14):2989-97. doi: 10.1113/jphysiol.2014.273995. Epub 2014 Apr 22. PMID 24756641
- [Background] Dinan TG, Cryan JF. Regulation of the stress response by the gut microbiota: implications for psychoneuroendocrinology. Psychoneuroendocrinology. 2012 Sep;37(9):1369-78. doi: 10.1016/j.psyneuen.2012.03.007. Epub 2012 Apr 5. PMID 22483040
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Bombardier C, Melfi CA, Paul J, Green R, Hawker G, Wright J, Coyte P. Comparison of a generic and a disease-specific measure of pain and physical function after knee replacement surgery. Med Care. 1995 Apr;33(4 Suppl):AS131-44. PMID 7723441
- [Background] Hawker G, Melfi C, Paul J, Green R, Bombardier C. Comparison of a generic (SF-36) and a disease specific (WOMAC) (Western Ontario and McMaster Universities Osteoarthritis Index) instrument in the measurement of outcomes after knee replacement surgery. J Rheumatol. 1995 Jun;22(6):1193-6. PMID 7674255
- [Background] McConnell S, Kolopack P, Davis AM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): a review of its utility and measurement properties. Arthritis Rheum. 2001 Oct;45(5):453-61. doi: 10.1002/1529-0131(200110)45:53.0.co;2-w. No abstract available. PMID 11642645
- [Background] Gill SD, de Morton NA, Mc Burney H. An investigation of the validity of six measures of physical function in people awaiting joint replacement surgery of the hip or knee. Clin Rehabil. 2012 Oct;26(10):945-51. doi: 10.1177/0269215511434993. Epub 2012 Feb 9. PMID 22324057
- [Background] Hill JC, Kang S, Benedetto E, Myers H, Blackburn S, Smith S, Dunn KM, Hay E, Rees J, Beard D, Glyn-Jones S, Barker K, Ellis B, Fitzpatrick R, Price A. Development and initial cohort validation of the Arthritis Research UK Musculoskeletal Health Questionnaire (MSK-HQ) for use across musculoskeletal care pathways. BMJ Open. 2016 Aug 5;6(8):e012331. doi: 10.1136/bmjopen-2016-012331. PMID 27496243
- [Background] Hill J, Kang S, Benedetto E, Myers H, Blackburn S, Smith S, et al. PMS74 - Development of the Musculoskeletal Health Questionnaire (MSK-HQ) for Use in Different Conditions and Different Healthcare Pathways. Value in Health. 2016;19(7):A544.
- [Background] Morley JE. Developing novel therapeutic approaches to frailty. Curr Pharm Des. 2009;15(29):3384-95. doi: 10.2174/138161209789105045. PMID 19860686
- [Background] Theou O, Stathokostas L, Roland KP, Jakobi JM, Patterson C, Vandervoort AA, Jones GR. The effectiveness of exercise interventions for the management of frailty: a systematic review. J Aging Res. 2011 Apr 4;2011:569194. doi: 10.4061/2011/569194. PMID 21584244
- [Background] Morley JE, Argiles JM, Evans WJ, Bhasin S, Cella D, Deutz NE, Doehner W, Fearon KC, Ferrucci L, Hellerstein MK, Kalantar-Zadeh K, Lochs H, MacDonald N, Mulligan K, Muscaritoli M, Ponikowski P, Posthauer ME, Rossi Fanelli F, Schambelan M, Schols AM, Schuster MW, Anker SD; Society for Sarcopenia, Cachexia, and Wasting Disease. Nutritional recommendations for the management of sarcopenia. J Am Med Dir Assoc. 2010 Jul;11(6):391-6. doi: 10.1016/j.jamda.2010.04.014. PMID 20627179
- [Background] Srinivas-Shankar U, Roberts SA, Connolly MJ, O'Connell MD, Adams JE, Oldham JA, Wu FC. Effects of testosterone on muscle strength, physical function, body composition, and quality of life in intermediate-frail and frail elderly men: a randomized, double-blind, placebo-controlled study. J Clin Endocrinol Metab. 2010 Feb;95(2):639-50. doi: 10.1210/jc.2009-1251. Epub 2010 Jan 8. PMID 20061435
- [Background] Morley JE, Malmstrom TK, Miller DK. A simple frailty questionnaire (FRAIL) predicts outcomes in middle aged African Americans. J Nutr Health Aging. 2012 Jul;16(7):601-8. doi: 10.1007/s12603-012-0084-2. PMID 22836700
- [Background] Bennell K, Dobson F, Hinman R. Measures of physical performance assessments: Self-Paced Walk Test (SPWT), Stair Climb Test (SCT), Six-Minute Walk Test (6MWT), Chair Stand Test (CST), Timed Up & Go (TUG), Sock Test, Lift and Carry Test (LCT), and Car Task. Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S350-70. doi: 10.1002/acr.20538. No abstract available. PMID 22588756
- [Background] Power JD, Perruccio AV, Badley EM. Pain as a mediator of sleep problems in arthritis and other chronic conditions. Arthritis Rheum. 2005 Dec 15;53(6):911-9. doi: 10.1002/art.21584. PMID 16342098
- [Background] Ancoli-Israel S. Sleep and its disorders in aging populations. Sleep Med. 2009 Sep;10 Suppl 1:S7-11. doi: 10.1016/j.sleep.2009.07.004. Epub 2009 Jul 31. PMID 19647483
- [Background] Senba E. A key to dissect the triad of insomnia, chronic pain, and depression. Neurosci Lett. 2015 Mar 4;589:197-9. doi: 10.1016/j.neulet.2015.01.012. Epub 2015 Jan 7. No abstract available. PMID 25576841
- [Background] Backhaus J, Junghanns K, Broocks A, Riemann D, Hohagen F. Test-retest reliability and validity of the Pittsburgh Sleep Quality Index in primary insomnia. J Psychosom Res. 2002 Sep;53(3):737-40. doi: 10.1016/s0022-3999(02)00330-6. PMID 12217446
- [Background] Akin-Akinyosoye K, Frowd N, Marshall L, Stocks J, Fernandes GS, Valdes A, McWilliams DF, Zhang W, Doherty M, Ferguson E, Walsh DA. Traits associated with central pain augmentation in the Knee Pain In the Community (KPIC) cohort. Pain. 2018 Jun;159(6):1035-1044. doi: 10.1097/j.pain.0000000000001183. PMID 29438225
- [Background] Broadbent DE, Cooper PF, FitzGerald P, Parkes KR. The Cognitive Failures Questionnaire (CFQ) and its correlates. Br J Clin Psychol. 1982 Feb;21(1):1-16. doi: 10.1111/j.2044-8260.1982.tb01421.x. PMID 7126941
- [Background] Bridger RS, Johnsen SA, Brasher K. Psychometric properties of the Cognitive Failures Questionnaire. Ergonomics. 2013;56(10):1515-24. doi: 10.1080/00140139.2013.821172. Epub 2013 Jul 23. PMID 23879800
- [Background] de Lange-Brokaar BJ, Ioan-Facsinay A, van Osch GJ, Zuurmond AM, Schoones J, Toes RE, Huizinga TW, Kloppenburg M. Synovial inflammation, immune cells and their cytokines in osteoarthritis: a review. Osteoarthritis Cartilage. 2012 Dec;20(12):1484-99. doi: 10.1016/j.joca.2012.08.027. Epub 2012 Sep 7. PMID 22960092
- [Background] Attur M, Samuels J, Krasnokutsky S, Abramson SB. Targeting the synovial tissue for treating osteoarthritis (OA): where is the evidence? Best Pract Res Clin Rheumatol. 2010 Feb;24(1):71-9. doi: 10.1016/j.berh.2009.08.011. PMID 20129201
- [Background] Guermazi A, Eckstein F, Hellio Le Graverand-Gastineau MP, Conaghan PG, Burstein D, Keen H, Roemer FW. Osteoarthritis: current role of imaging. Med Clin North Am. 2009 Jan;93(1):101-26, xi. doi: 10.1016/j.mcna.2008.08.003. PMID 19059024
- [Background] Sarmanova A, Hall M, Moses J, Doherty M, Zhang W. Synovial changes detected by ultrasound in people with knee osteoarthritis - a meta-analysis of observational studies. Osteoarthritis Cartilage. 2016 Aug;24(8):1376-83. doi: 10.1016/j.joca.2016.03.004. Epub 2016 Mar 10. PMID 26973325
- [Background] Snelling SJ, Bas S, Puskas GJ, Dakin SG, Suva D, Finckh A, Gabay C, Hoffmeyer P, Carr AJ, Lubbeke A. Presence of IL-17 in synovial fluid identifies a potential inflammatory osteoarthritic phenotype. PLoS One. 2017 Apr 11;12(4):e0175109. doi: 10.1371/journal.pone.0175109. eCollection 2017. PMID 28399156
- [Background] Berkoff DJ, Miller LE, Block JE. Clinical utility of ultrasound guidance for intra-articular knee injections: a review. Clin Interv Aging. 2012;7:89-95. doi: 10.2147/CIA.S29265. Epub 2012 Mar 20. PMID 22500117
- [Background] Haavardsholm EA, Aga AB, Olsen IC, Lillegraven S, Hammer HB, Uhlig T, Fremstad H, Madland TM, Lexberg AS, Haukeland H, Rodevand E, Hoili C, Stray H, Noraas A, Hansen IJ, Bakland G, Nordberg LB, van der Heijde D, Kvien TK. Ultrasound in management of rheumatoid arthritis: ARCTIC randomised controlled strategy trial. BMJ. 2016 Aug 16;354:i4205. doi: 10.1136/bmj.i4205. PMID 27530741
- [Background] Sibbitt WL Jr, Kettwich LG, Band PA, Chavez-Chiang NR, DeLea SL, Haseler LJ, Bankhurst AD. Does ultrasound guidance improve the outcomes of arthrocentesis and corticosteroid injection of the knee? Scand J Rheumatol. 2012 Feb;41(1):66-72. doi: 10.3109/03009742.2011.599071. Epub 2011 Nov 21. PMID 22103390
- [Background] Palmieri-Smith RM, Thomas AC, Karvonen-Gutierrez C, Sowers MF. Isometric quadriceps strength in women with mild, moderate, and severe knee osteoarthritis. Am J Phys Med Rehabil. 2010 Jul;89(7):541-8. doi: 10.1097/PHM.0b013e3181ddd5c3. PMID 20463561
- [Background] Tan J, Balci N, Sepici V, Gener FA. Isokinetic and isometric strength in osteoarthrosis of the knee. A comparative study with healthy women. Am J Phys Med Rehabil. 1995 Sep-Oct;74(5):364-9. PMID 7576413
- [Background] Berry PA, Jones SW, Cicuttini FM, Wluka AE, Maciewicz RA. Temporal relationship between serum adipokines, biomarkers of bone and cartilage turnover, and cartilage volume loss in a population with clinical knee osteoarthritis. Arthritis Rheum. 2011 Mar;63(3):700-7. doi: 10.1002/art.30182. PMID 21305502
- [Background] Richette P, Poitou C, Garnero P, Vicaut E, Bouillot JL, Lacorte JM, Basdevant A, Clement K, Bardin T, Chevalier X. Benefits of massive weight loss on symptoms, systemic inflammation and cartilage turnover in obese patients with knee osteoarthritis. Ann Rheum Dis. 2011 Jan;70(1):139-44. doi: 10.1136/ard.2010.134015. Epub 2010 Oct 26. PMID 20980288
- [Background] Mouritzen U, Christgau S, Lehmann HJ, Tanko LB, Christiansen C. Cartilage turnover assessed with a newly developed assay measuring collagen type II degradation products: influence of age, sex, menopause, hormone replacement therapy, and body mass index. Ann Rheum Dis. 2003 Apr;62(4):332-6. doi: 10.1136/ard.62.4.332. PMID 12634232
- [Background] Duvall MG, Levy BD. DHA- and EPA-derived resolvins, protectins, and maresins in airway inflammation. Eur J Pharmacol. 2016 Aug 15;785:144-155. doi: 10.1016/j.ejphar.2015.11.001. Epub 2015 Nov 3. PMID 26546247

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Started | 14 | 57
Completed | 14 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation | Total
Number analyzed (Participants) | 11 | 46 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 15 | 19
  >=65 years | 7 | 31 | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (6.5) | 68.7 (6.5) | 66.9 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 20 | 27
  Male | 4 | 26 | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 11 | 46 | 57

OUTCOME MEASURES:

1. Primary Outcome: Pain Sensitivity: Pressure Pain Detection Threshold (PPT)
Description: PPT is a non-invasive test during which the sensitivity of the nerves is assessed by recording the amount of pressure applied to the skin. Pressure is applied through a probe. The pressure probe used is mounted in a handheld device connected to a computer. Pressure applied to the skin is gradually increased until the participant indicates (by pressing a button) that the sensation has changed from pressure to pain. The probe will be used on the contralateral forearm (brachioradialis muscle) using a standardised protocol used in other studies within the Pain Centre. Each region will be tested one time with short rest periods between each. The participants will be familiarised with the test before it is administered so that they know what to expect and how to respond.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
kPa | 252.58 (124.41) | 266.17 (93.82)

2. Primary Outcome: Pain Sensitivity: Temporal Summation Pain (TS)
Description: TS is a non-invasive test during which repetitive mechanical stimulation is applied over a short period to get their augmented response. A 256mN weighted pinprick stimulator will be used and applied perpendicular to the skin of suprapatellar region of the painful knee (5cm proximal from the centre of patella). The participant will be asked to rate the pain or sharpness they experience from 0-10 where 0 indicates no pain or sharpness and 10 indicates the most intense pain or sharpness imaginable. The response of the participant will be recorded. The same stimulator at the same site will be applied ten times repeatedly at a rate of 1/second. At the end of the series of 10 pinpricks, the participant will be asked to rate the average pain or sharpness they experienced out of the 10 stimuli using the same scale. The TS value will be calculated as the difference between the two ratings (single stimulus minus the average of the 10 stimuli).
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale | 4.26 (0.71) | 0.91 (0.83)

3. Primary Outcome: Pain Sensitivity: Conditioned Pain Modulation (CPM)
Description: CPM is the application of PPT before and while a pressure cuff is inflated. A 7.5cm wide tourniquet cuff will be wrapped around the arm contra-laterally to the most painful knee. The lower rim of tourniquet cuff will be kept 3cm proximal to cubital fossa. The cuff will be inflated with the aim to reach above-systolic pressure with a maximum of 270mm/Hg. After target pressure is achieved, the participant will be asked to repeatedly make a handgrip or squeeze a foam ball until they develop ischemic pain ≥4 out of 10 on a 0-10 scale. Once NRS of 4/10 will be achieved, the probe of algometer will be applied in the same manner as during PPT testing. Once the participant presses the button, the probe will be withdrawn, and the cuff will be deflated released from the participants arm. The difference in PPT score (PPT with conditioning minus PPT without conditioning) will be considered the CPM value. A positive value indicates efficient CPM whereas a negative value indicates impaired CPM.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: kPa
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
kPa | 73.66 (92.05) | 13.85 (137.71)

4. Secondary Outcome: Central Aspects of Knee Pain (CAP-Knee)
Description: Central augmented pain assessed on a 8-item CAP-Knee questionnaire, where items 1-7 are scored from 0-3, 0 indicating "never" and 3 indicating "often" or "always". Item 8 (pain distribution manikin) was allocated a score of 0 if at most 1 knee is shades, and no other regions below the waist, or a score of 3 if both knees were shaded, or one knee plus any additional shaded areas below the waist. A total sum score (minimum score of "0", maximum score of "24") will be calculated for analysis. The higher the value the higher the levels of central augmented pain.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Non-prevalent Central Sensitisation: All other participants with sensitisation that is not significantly deviating from the normal mean as assessed by Quantitative Sensory Testing
  Q
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
Score on a scale | 8.9 (3.4) | 6.2 (2.4)

5. Secondary Outcome: Anxiety
Description: Anxiety will be assessed with the Anxiety part of the Hospital Anxiety and Depression Scale (HADS) where patients are asked to indicate their levels of emotion frequency with a 4-level scale (0-3: 0 indicates never and 3 all the time) at 7 questions. A sum of all responses is calculated (minimum score of "0", maximum score of "21") for analysis. The higher the value the higher the levels of anxiety.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale | 6.00 (3.67) | 5.56 (2.94)

6. Secondary Outcome: Depression
Description: Depression will be assessed with the Depression part of the Hospital Anxiety and Depression Scale (HADS) where patients are asked to indicate their levels of emotion frequency with a 4-level scale (0-3: 0 indicates all the time and 3 never) at 7 questions. A sum of all responses is calculated (minimum score of "0", maximum score of "21") for analysis. The higher the value the higher the levels of depression.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale | 4.00 (3.12) | 5.15 (2.74)

7. Secondary Outcome: Cognitive Function
Description: Cognitive function will be assessed with the Cognitive Failures Questionnaire (CFQ) where participants are asked to indicate symptom frequency with a 0-4 scale (0 indicates never and 4 very often) on 25 statements. A sum of all responses is calculated (minimum score of "0", maximum score of "100") for analysis. The higher the value the more impaired cognitive function is.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale | 36.7 (14.8) | 35.8 (11.4)

8. Secondary Outcome: Sleep Quality
Description: Sleep quality will be assessed with the Pittsburgh Sleep Quality Index (PSQI) where participants are asked to respond to 18 statements indicating their: 1) sleep duration in minutes/hours on 4 questions, 2) symptom frequency with 4 possible answers spreading from 'not during the past month' to 'three or more times a week' on 12 statements, 3) symptom severity with 4 possible answers spreading from 'no problem at all' to 'very big problem' on 1 statement and 4) sleep quality with 4 possible answers spreading from 'very good' to 'very bad' on 1 statement. Responses are coded from 0-4 (0 indicating no sleeping issues and 4 frequent and severe sleeping problems). A sum of all 18 responses is calculated (minimum score of "0", maximum score of "72" being the maximum) for analysis. The higher the value the less sleep quality there is.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale | 1.22 (0.44) | 1.27 (0.78)

9. Secondary Outcome: Knee Pain, Stiffness, and Physical Functioning
Description: Knee pain, stiffness and physical functioning will be assessed with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) where participants are asked to rate their symptom severity with a 0-4 scale (0 indicates never and 4 extreme) five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). The higher the value in each domain the more pain, stiffness and physical dysfunction there is.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale
  Physical Function | 31.00 (15.23) | 27.07 (11.78)
  Stiffness | 4.44 (1.67) | 4.17 (1.49)
  Pain | 9.44 (3.91) | 8.10 (3.37)

10. Secondary Outcome: General Musculoskeletal Health
Description: General health will be assessed with the Musculoskeletal Health Questionnaire (MSK-HQ) where participants are asked to indicate symptom frequency with a 0-4 scale (0 indicates very severe and 4 not at all severe) on 14 statements. A sum of all responses is calculated (minimum score of "0", maximum score of "56") for analysis. The lower the value the more reduced general musculoskeletal health is.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale | 4.44 (2.24) | 2.73 (2.23)

11. Secondary Outcome: Frailty
Description: Frailty will be measured with a modified questionnaire where participants will be asked to respond to 8 Yes/No questions (Yes is marked with 1 and No with 0) about inability to walk, using aids, weight loss, co-morbidities and levels of physical activity. A total out of all responses (minimum score of "0", maximum score of "8") is calculated for analysis. The higher the score, the higher the levels of frailty
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 11 | 46
score on a scale | 1.33 (1.50) | 1.07 (1.20)

12. Other Pre Specified Outcome: Dietary Habits (OPTIONAL)
Description: Dietary habits will be assessed with the Food Frequency Questionnaire (FFQ) where participants are asked to indicate the consumption frequency of different types of food materials with a 0-9 scale (0 indicates 'never or less than once a month' and 9 'more than 6 times per day') on 150 distinct foods divided into dairy, fruits, vegetables, meat and fish, soups, bread, sweets, potatoes, and beverages. A total score is calculated for each category with the maximum depending on the amount of items in each category. The larger the total value the more frequent the consumption of a food category per day is.
Time Frame: At baseline
Population: Not enough questionnaires were returned to allow for meaningful statistical analysis
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
Number analyzed (Participants) | 0 | 0

13. Other Pre Specified Outcome: Biosamples (Synovial Fluid A)
Description: Concentration of inflammatory markers (cytokines) identified in extracted synovial fluid.
Time Frame: At baseline
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Biosamples (Synovial Fluid B)
Description: Concentration of proteomic concentrations (fibronectin) identified in extracted synovial fluid.
Time Frame: At baseline
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Biosamples (Synovial Fluid C)
Description: Concentration of gene expression molecules (RNA polymerase II) identified in extracted synovial fluid.
Time Frame: At baseline
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Biosamples (Blood A)
Description: Concentration of stress markers (cortisol) identified in participants' blood samples.
Time Frame: At baseline
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Biosamples (Blood B)
Description: Concentration of insulin resistance markers (fasting blood glucose) identified in participants' blood samples.
Time Frame: At baseline
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Biosamples (Blood C)
Description: Concentration of metabolic rate markers (triglycerides) identified in participants' blood samples.
Time Frame: At baseline
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Biosamples (Urine A)
Description: Concentration of metabolic rate markers (UTXII collagen degradation marker) identified in participants' urine samples.
Time Frame: At baseline
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Biosamples (Urine B)
Description: Concentration of inflammatory regulator markers (maresins) identified in participants' urine samples.
Time Frame: At baseline
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Biosamples (Saliva)
Description: Concentration of stress markers (cortisol) in participants' saliva samples.
Time Frame: At baseline
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Biosamples (Faeces A) [OPTIONAL]
Description: Concentration of metabolic rate markers (glucosamine) in participants' faecal samples.
Time Frame: At baseline
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Biosamples (Faeces B) [OPTIONAL]
Description: Concentration of metabolic rate markers (chondroitin sulfate) in participants' faecal samples.
Time Frame: At baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: At baseline session, throughout the session. No monitoring took place after the end of the baseline session
Description: 57 people. No adverse event were reported after systematic assessment.
Arm/Group | Prevalent Central Sensitisation | Non-prevalent Central Sensitisation
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/46
Other Adverse Events (participants affected / at risk) | 0/11 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT04443452/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT04443452/ICF_000.pdf